CLINICAL TRIAL: NCT05374460
Title: Factors Affecting Sensory and Motor Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hannah Justine Block, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14804; R01NS112367-01A1 (NIH)
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Basic Science

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Conscious awareness: No information (Sham Comparator): Told nothing about the visuo-proprioceptive mismatch. Hand remains hidden beneath mirror that shows visual display. (control)
  Interventions: Behavioral: Attend to the targets
- Conscious awareness: Explanatory diagram (Experimental): Told in advance about the visuo-proprioceptive mismatch, which will be explained with a diagram. Hand remains hidden.
  Interventions: Behavioral: Explanatory diagram
- Conscious awareness: Direct vision of hand (Experimental): Foamboard under mirror removed, making the mirror see-through and the hand directly visible.
  Interventions: Behavioral: Direct vision
- Movement feedback: No feedback (Sham Comparator): No movement feedback (control)
  Interventions: Behavioral: No movement feedback
- Movement feedback: Target hand (Experimental): Movement feedback about the target hand.
  Interventions: Behavioral: Movement feedback, target hand
- Movement feedback: Pointing hand (Experimental): Movement feedback about the pointing hand.
  Interventions: Behavioral: Movement feedback, pointing hand

INTERVENTIONS:
Behavioral: Explanatory diagram — Participant is told there will be a mismatch between their target finger and the visual indicator of target finger position. They will be shown a diagram explaining this.
  Arms: Conscious awareness: Explanatory diagram
Behavioral: Direct vision — Foamboard under mirror removed, making the mirror see-through and the hand directly visible. Mismatch between target hand and visual indicator will be directly visible.
  Arms: Conscious awareness: Direct vision of hand
Behavioral: Movement feedback, target hand — After the participant points at each target, a cursor indicating final pointing position will be displayed briefly. The visual indicator of the target hand will be displaced.
  Arms: Movement feedback: Target hand
Behavioral: Movement feedback, pointing hand — After the participant points at each target, a cursor indicating final pointing position will be displayed briefly. The visual indicator of the target hand will not change, but the cursor indicating pointing hand position will change.
  Arms: Movement feedback: Pointing hand
Behavioral: No movement feedback — The visual indicator of the target hand will be displaced, but there will be no cursor to indicate the pointing hand's position.
  Arms: Movement feedback: No feedback
Behavioral: Attend to the targets — Participants will not be told anything about the visuo-proprioceptive mismatch. Instead, they will be asked simply to attend to the target positions.
  Arms: Conscious awareness: No information

SUMMARY:
How participants perceive the position of their own hand in various contexts will be examined. This will include changing the visual display to suggest the hand is in a slightly different position, and asking participants to indicate where they think it is by pointing with their other hand.

DETAILED DESCRIPTION:
Hand position can be estimated visually, from an image on the retina, and proprioceptively, from sensors in the joints, muscles, and skin. The brain is thought to weight and combine available sensory estimates to form an integrated multisensory estimate. Inherent in this process is the capacity to realign one or both sensory estimates when they become spatially mismatched, as when washing dishes with the hands immersed in water, which refracts light. It is generally assumed that if a person knows about the sensory mismatch somehow, the realignment will not occur. This assumption will be tested in two experiments by giving people this information in different ways. Expt. A: Conscious awareness of the mismatch will be presented in different ways, or absent. Expt. B: Movement error feedback will be presented in different ways, or absent.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45 years old
* Right-handed.
* Covid has been found to have neurological effects in some people, but mostly the effects on sensorimotor control and neurophysiology are unknown. So we will only include individuals who report being free of Covid symptoms in week preceding testing.

Exclusion Criteria:

* Past or present history of seizure, stroke, any brain or peripheral nerve disease, severe head trauma, or spinal cord surgery.
* Learning or attention conditions such as ADHD.
* Orthopedic or pain conditions, or a history of seriously injured bones, joints or muscles in either arm.
* Lack of normal or corrected-to-normal vision.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Realignment | 1 day
  Measured by comparing where the subject points on a touchscreen when indicating perceived position of visual and proprioceptive targets early vs. late in the behavioral task.

SECONDARY OUTCOMES:
Visuo-proprioceptive weighting | 1 day
  The degree to which participant relies on vision vs. proprioception when both are available. Measured by comparing where the subject points on a touchscreen when indicating perceived position of visual vs. proprioceptive targets.
Target estimation variance | 1 day.
  Variance with which participant estimate visual and proprioceptive target positions. Computed from where subjects point at targets on a touchscreen.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah J Block, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Hannah Block, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results published in peer-reviewed journals will be shared. Only de-identified data will be shared.
Supporting Information: Analytic Code
Time Frame: The data will become available when group results are published in peer-reviewed journals.
Access Criteria: Data will be available on www.osf.io for anyone who wishes to download it. The relevant osf registry will be cited in the peer-reviewed publication so that interested readers can find it.